CLINICAL TRIAL: NCT00310596
Title: Cardiovascular Safety Study of 0.1 and 0.3 mmol/kg Magnevist® Injection at Two Injection Rates (Bolus and 10 mL/15 Sec.) in Normal Subjects Following a Randomized, Cross-over Design Using Placebo and a Concurrent Positive Control
Brief Title: Cardiovascular Safety Study of Magnevist® Injection at Two Dose Levels and Two Injection Rates in Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 91024; 305340
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: ECG safety
MeSH Terms: interventions — Gadolinium DTPA; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)
- Arm 2 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)
- Arm 3 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)
- Arm 4 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)
- Arm 5 (Active Comparator)
  Interventions: Drug: Moxifloxacin (BAY12-8039)
- Arm 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — 0,1mmol/kg at 10 mL/15 sec
  Arms: Arm 1
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — same dose as arm 1 at bolus rate (2mL/sec)
  Arms: Arm 2
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — 0,3mmol/kg at 10 mL/15 sec
  Arms: Arm 3
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — same dose as arm 3 at bolus rate (2mL/sec)
  Arms: Arm 4
Drug: Moxifloxacin (BAY12-8039) — 400 mg at 0,07 mL/sec over 60 min
  Arms: Arm 5
Drug: Placebo — 0,9% saline at 0,6mL/kg at bolus rate
  Arms: Arm 6

SUMMARY:
The purpose of this study is to determine what effect Magnevist (gadopentetate dimeglumine) injection has on the way the heart conducts the electrical impulses that allow it to beat effectively. The study will compare Magnevist injection's effect to that of placebo (a saline injection).

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an electrocardiogram [ECG] (normal sinus rhythm [SR], QTc > 450 msec) without clinically significant abnormalities
* Non-smoker

Exclusion Criteria:

* History of cardiovascular disease- Pregnant or nursing- Had any contraindication to moxifloxacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2004-01; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
The primary study variable was heart-rate corrected QT (QTc) interval | Within 15 min postinjection

SECONDARY OUTCOMES:
Adverse event monitoring, laboratory evaluations | 24 hrs postinjection
ECG variables and overall interpretation | 24 hrs postinjection

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Miami, Florida, United States